CLINICAL TRIAL: NCT05004545
Title: To Compare Hemodynamic Parameters of Propofol and Sevoflurane During Cardiopulmonary Bypass Time in Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery to Avoid Lactate Level.
Brief Title: Compare Hemodynamic Parameters of Propofol and Sevoflurane During CPB Time in Undergoing CABG to Avoid Lactate Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaudhry Pervaiz Elahi Institute of Cardiology (Other Government)
Responsible Party: Principal Investigator, Muhammad Imran Khan, Principal investigator, Chaudhry Pervaiz Elahi Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CPEIC-06
Record Dates: First submitted 2021-07-16; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Hemodynamic Instability
Keywords: Propofol; Sevoflurane; hemodynamic stability; Lactate level
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 Profol Infusion to CABG patients to check lactate level (Experimental): Propofol infusion according to bodyweight will be given to check lactate level on CPB
  Interventions: Drug: Propofol
- sevoflurane will be given to group 2 to check lacate level (Active Comparator): Sevoflurane MAC % will be given to CABG patients to check lactate level
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol infusion according to body weight will be compared with sevoflurane acording to MAC % to see the lactate level and hemodynamic parameters of CABG patients

SUMMARY:
Hemodynamic parameters and lactate level will be on CBP during CABG surgery patients.

DETAILED DESCRIPTION:
Objective: To compare hemodynamic parameters of propofol and sevoflurane during cardiopulmonary bypass time in patients undergoing coronary artery bypass graft (CABG) surgery to avoid lactate level.

Methods: One hundred and twenty six patients scheduled for CABG from May 2017 to May 2018 will be included in this study. Non probability consecutive sampling will be used. Patients will be divided in two groups, propofol will be given to group 1, and sevoflurane will be given to group 2. Age, clamp time, bypass time, mean arterial blood pressure on bypass machine and lactate level will be compared between two groups. SPSS version 24 will used and p value ≤ 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

CABG

Exclusion Criteria:

Emergency surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-06-10 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Lactate level will be measured during CPB for CABG patients to see the hemodynamics parameters | 06 months
  The mean pre-cross clamp lactate level and post- rewarming lactate level will be calculated to see the effect of this on the CABG patients hemodynamics during CBP

CONTACTS AND LOCATIONS:
Overall Officials: Kaneez Ume Farwa, FCPS, Principal Investigator — Chaudhry Pervaiz Elahi Institute of Cardiology
Locations (1):
- Cardiac Surgery ICU, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Ok
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Soon
Access Criteria: Ok